CLINICAL TRIAL: NCT03106961
Title: An Optical Coherence Tomography Evaluation of the Effects of High-Pressure, Non-compliant Ballooning on Scaffold Embedding
Brief Title: OCT and Scaffold Embedding After NC Balloon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Francis Hospital, New York (Other)
Collaborators: Akiko Maehara, MD (Unknown)
Responsible Party: Principal Investigator, Richard A. Shlofmitz, MD, Chairman of Cardiology, St. Francis Hospital, New York
Other Study IDs: 16-19
Record Dates: First submitted 2016-10-04; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bioresorbable vascular scaffolds, OCT, non-compliant ballooning — Measure the effect of high-pressure, NC ballooning on scaffold embedding by OCT

SUMMARY:
This study is a single-center, prospective, observational study designed to subjects presenting with stable angina pectoris or acute coronary syndromes requiring treatment of de novo lesions.

Eligible subjects will have BVS scaffold implant using a high pressure post-scaffold implantation ballooning, designed to specifically address the issue of incomplete BVS expansion. OCT ( optical coherence tomography ) will be used to evaluate the change in the intraluminal scaffold volume and the prevalence of scaffold embedding from post-scaffold implantation to post-dilation high pressure (16-20 atm), non-compliant ballooning in relation to the underlying plaque.

DETAILED DESCRIPTION:
This study is a single-center, prospective, observational study designed to enroll 50 subjects presenting with stable angina pectoris or acute coronary syndromes requiring treatment of de novo lesions. Consented subjects are to undergo PCI and have a lesion without angiographic calcification.

Eligible subjects who meet inclusion and exclusion criteria for BVS scaffold implant will have a BVS-specific implantation protocol with high pressure post-scaffold implantation ballooning, designed to specifically address the issue of incomplete BVS expansion. Because the scaffold is compliant, a perfectly embedded scaffold is sometimes observed in a lesion with soft plaque, resulting in a smaller intra-luminal scaffold volume that may reduce the event rate. Enrolled subjects will have OCT ( optical coherence tomography ) pre and post BVS implantation to assess the change in the intraluminal scaffold volume and the prevalence of scaffold embedding from post-scaffold implantation (using the moderate pressure of 12 atm) to post-dilation high pressure (16-20 atm), non-compliant ballooning in relation to the underlying plaque.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years who undergo PCI of de novo lesions in the setting of stable angina or acute coronary syndromes.
2. The culprit lesion must be successfully pre-dilated prior to enrollment. -

Exclusion Criteria:

I. Patient specific

1. Cardiogenic shock (sustained [>10 min] systolic blood pressure <90 mm Hg in absence of inotropic support or the presence of an intra-aortic balloon pump support).
2. Known severe renal insufficiency (estimated glomerular filtration rate <30 mL/min/1.72 m2).
3. Intolerance of aspirin or thienopyridines
4. ST-segment elevation myocardial infarction
5. Subject is a woman of childbearing potential, pregnant, or nursing.
6. Subject has received a heart transplant or any other organ transplant or is on a waiting list for any organ transplant.
7. Subject has a known hypersensitivity or contraindication to aspirin, both heparin and bivalirudin, clopidogrel, ticlopidine, ticagrelor or prasugrel, or to everolimus, PLLA polymers, or contrast sensitivity that cannot be adequately pre-medicated.
8. Subject has a platelet count <100,000 cell/mm3 or >700,000 cell/mm3, a white blood cell count of <3,000 cell/mm3, or documented or suspected liver disease in the recent blood test.

II. Lesion specific

1. Left main disease defined as diameter stenosis >50%
2. Ostial lesion
3. Tortuous artery in which OCT is unable to pass
4. Lesion in a bypass graft
5. Reference vessel diameter (RVD) <2.5 mm or >4 mm
6. Bifurcation lesions with side branches >2 mm
7. In-stent restenosis
8. Previous placement of a stent proximal or distal to or within 10 mm of the target lesion
9. Chronic total occlusion
10. Lesions with calcified plaque >180° by pre-intervention OCT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 50 subjects presenting with stable angina pectoris or acute coronary syndromes requiring treatment of de novo lesions. Consented subjects are to undergo PCI and have a lesion without angiographic calcification.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-03-22 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of the number of embedded scaffold struts as evaluated by OCT | intra-procedure (PCI)
  Percentage of embedded scaffold strut is defined as the ratio of the number of embedded strut to the total number of analyzed strut per lesion. (% of embedded scaffold struts = No. of embedded struts / total No. of analyzed struts) The analysis will be done for both OCT images 1) after initial bioresorbable scaffold implantation using moderate pressure and 2) after post-dilatation using high pressure non-compliant balloon, and the change in percentage of embedded scaffold strut from initial bioresorbable scaffold implantation to post-dilation will be calculated. (∆ % of embedded scaffold struts = % of embedded scaffold struts of initial scaffold implantation - % of embedded scaffold struts of post-dilatation)

SECONDARY OUTCOMES:
Change in minimum scaffold cross-sectional area | intra-procedure (PCI)
  Minimum scaffold cross-sectional area defined as the smallest endoluminal area within the entire scaffold cross-section. We will evaluate the change from initial bioresorbable scaffold implantation using moderate pressure to post-dilation using high pressure using non-compliant balloon
Change in mean scaffold cross-sectional area | intra-procedure (PCI)
  Mean scaffold cross-sectional area defined as the average of endoluminal area within the entire scaffold cross-section. We will evaluate the change from initial bioresorbable scaffold implantation using moderate pressure to post-dilation using high pressure using non-compliant balloon
Change in the ratio of minimum scaffold cross-sectional area and expected scaffold cross-sectional area from manufacturer chart of balloon | intra-procedure (PCI)
  We will evaluate the change from initial bioresorbable scaffold implantation using moderate pressure to post-dilation using high pressure using non-compliant balloon.
Change in the ratio of minimum scaffold cross-sectional area and average of proximal and distal reference lumen cross-sectional | intra-procedure (PCI)
  We will evaluate the change from initial bioresorbable scaffold implantation using moderate pressure to post-dilation using high pressure using non-compliant balloon
Change in the Percentage of footprint | intra-procedure (PCI)
  Percentage of footprint defined as the ratio of outer BVS scaffold surface area to total luminal surface area. We will evaluate the change from initial bioresorbable scaffold implantation using moderate pressure to post-dilation using high pressure using non-compliant balloon
Comparison of scaffold embedding between non-calcified plaque and moderate calcified plaque (arc <180°) | intra-procedure (PCI)
  In the strut level, the percentage of embedded scaffold struts between calcified plaque and non-calcified plaque will be compared. And about the lesion, Other secondary endpoints(2-7) listed above will be compared between calcified plaque and non-calcified plaque will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Shlofmitz, MD, Principal Investigator — St FrancisHospiral
Locations (1):
- St Francis Hospital, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Capodanno D, Gori T, Nef H, Latib A, Mehilli J, Lesiak M, Caramanno G, Naber C, Di Mario C, Colombo A, Capranzano P, Wiebe J, Araszkiewicz A, Geraci S, Pyxaras S, Mattesini A, Naganuma T, Munzel T, Tamburino C. Percutaneous coronary intervention with everolimus-eluting bioresorbable vascular scaffolds in routine clinical practice: early and midterm outcomes from the European multicentre GHOST-EU registry. EuroIntervention. 2015 Feb;10(10):1144-53. doi: 10.4244/EIJY14M07_11. PMID 25042421
- [Background] Brugaletta S, Gori T, Low AF, Tousek P, Pinar E, Gomez-Lara J, Scalone G, Schulz E, Chan MY, Kocka V, Hurtado J, Gomez-Hospital JA, Munzel T, Lee CH, Cequier A, Valdes M, Widimsky P, Serruys PW, Sabate M. Absorb bioresorbable vascular scaffold versus everolimus-eluting metallic stent in ST-segment elevation myocardial infarction: 1-year results of a propensity score matching comparison: the BVS-EXAMINATION Study (bioresorbable vascular scaffold-a clinical evaluation of everolimus eluting coronary stents in the treatment of patients with ST-segment elevation myocardial infarction). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt B):189-197. doi: 10.1016/j.jcin.2014.10.005. PMID 25616924
- [Background] Stone GW, Gao R, Kimura T, Kereiakes DJ, Ellis SG, Onuma Y, Cheong WF, Jones-McMeans J, Su X, Zhang Z, Serruys PW. 1-year outcomes with the Absorb bioresorbable scaffold in patients with coronary artery disease: a patient-level, pooled meta-analysis. Lancet. 2016 Mar 26;387(10025):1277-89. doi: 10.1016/S0140-6736(15)01039-9. Epub 2016 Jan 27. PMID 26825231
- [Background] Cassese S, Byrne RA, Ndrepepa G, Kufner S, Wiebe J, Repp J, Schunkert H, Fusaro M, Kimura T, Kastrati A. Everolimus-eluting bioresorbable vascular scaffolds versus everolimus-eluting metallic stents: a meta-analysis of randomised controlled trials. Lancet. 2016 Feb 6;387(10018):537-544. doi: 10.1016/S0140-6736(15)00979-4. Epub 2015 Nov 17. PMID 26597771
- [Background] Puricel S, Cuculi F, Weissner M, Schmermund A, Jamshidi P, Nyffenegger T, Binder H, Eggebrecht H, Munzel T, Cook S, Gori T. Bioresorbable Coronary Scaffold Thrombosis: Multicenter Comprehensive Analysis of Clinical Presentation, Mechanisms, and Predictors. J Am Coll Cardiol. 2016 Mar 1;67(8):921-931. doi: 10.1016/j.jacc.2015.12.019. PMID 26916481